CLINICAL TRIAL: NCT03251521
Title: Evaluation of Pain Intensity in Different Steps of Injection With Botulinum Toxin in the Treatment of Spasticity in Post-stroke Patients
Brief Title: Pain During Injection With Botulinum Toxin in Post-stroke Spasticity Treatment
Acronym: DOLOTOX
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC17.251
Record Dates: First submitted 2017-08-11; First posted 2017-08-16 (Actual); Last update posted 2017-08-16 (Actual); Status verified 2017-08

CONDITIONS: Post-stroke Spasticity
Keywords: pain; spasticity; stroke; injection; botulinum toxin A
MeSH Terms: conditions — Pain; Muscle Spasticity; Stroke | interventions — Botulinum Toxins

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- spasticity post-stroke: pain rating during injection with botulinum toxin The pain intensity was rated verbally on a numeric scale
  Interventions: Other: pain rating during injection with botulinum toxin

INTERVENTIONS:
Other: pain rating during injection with botulinum toxin — The pain intensity was rated verbally on a numeric scale. The pain was rated after each phase of injection

SUMMARY:
The aim of the study was to analyze which step of the procedure of toxin botulinum injection is the most painful between skin break-in, electric stimulation, injection and needle withdrawal.

DETAILED DESCRIPTION:
Post-stroke spasticity management by botulinum toxin injections may be limited by pain or discomfort at the injection side.

Particularly tracking by electrostimulation, but also skin puncture, toxin injection or needle withdrawal may be painful.

The objective of this study is to define an individual injection strategy in order to limit pain.

ELIGIBILITY:
Inclusion Criteria:

* stroke
* severe upper or lower limb spasticity (Ashworth score ≥ 2 for at least one muscle)
* patients requiring a treatment by botulinum toxin
* patients refusing analgesia for injections.

Exclusion Criteria:

* severe aphasia (severity subscore of the BDAE <3)
* cognitive impairment or psychiatric disease altering the reliability of pain evaluation
* patient medically unstable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients were assessed during routine botulinum toxin injection in the day clinic of our department
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Evolution of pain intensity during injection with botulinum toxin | 30 min
  Pain intensity in different steps of the procedure of toxin botulinum injection: skin break-in, electric stimulation, injection and needle withdrawal.

SECONDARY OUTCOMES:
Hypoesthesia | 30 min
  Semmes Weinstein Monofilament Evaluation
Neuropathic pain | 30 min
  DN4 (Neuropathic pain 4 questions)

CONTACTS AND LOCATIONS:
Overall Officials: Dominic PERENNOU, MD, PhD, Principal Investigator — University Hospital, Grenoble

IPD SHARING:
Plan to Share IPD: No